CLINICAL TRIAL: NCT00147823
Title: A Prospective Randomized Study Comparing Vitoss Alone Versus Vitoss With Bone Marrow Aspirate in Benign Bone Lesions
Brief Title: Comparing Synthetic Bone Alone Versus Synthetic Bone With Bone Marrow in Bone Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Orthovita d/b/a Stryker (Industry)
Responsible Party: Principal Investigator, Timothy Damron, M.D., Associate Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUNY UMU IRB # 5130
Record Dates: First submitted 2005-09-01; First posted 2005-09-07 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2013-12

CONDITIONS: Bone Diseases
Keywords: Bone formation; Bone lesions; Benign bone lesion
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitoss with bone marrow aspirate (Experimental): Addition of Vitoss to the bone marrow aspirate
  Interventions: Device: Vitoss with Bone Marrow Aspirate
- Vitoss Alone (Active Comparator): vitoss alone
  Interventions: Device: Vitoss Alone

INTERVENTIONS:
Device: Vitoss Alone — Synthetic bone graft material
  Arms: Vitoss Alone
Device: Vitoss with Bone Marrow Aspirate — Vitoss mixed with Bone Marrow aspirate
  Arms: Vitoss with bone marrow aspirate

SUMMARY:
This is a prospective randomized study comparing Vitoss alone versus Vitoss with bone marrow aspirate in benign bone lesions.

DETAILED DESCRIPTION:
Bone graft obtained from a patient's own bone (autogenous), usually around the pelvis, is currently considered the gold standard for bone grafting material. It provides a structural scaffold on which the patient's own bone may grow into (osteoconduction), growth factors that can stimulate healing (osteoinduction), and primitive cells (progenitors) that can stimulate bone formation directly (osteogenesis). It readily regains a blood supply from the surrounding tissues (revascularization) and is incorporated into the recipient site. However, there are significant disadvantages in the use of the patient's own bone graft including complications where the bone is taken from (donor site morbidity), limited availability and expense. For defects created by scraping (curettage) of non-cancerous (benign) bone lesions, a structural scaffold (osteoconduction) is generally considered the minimal necessary role that the graft material must serve to allow healing of the defect. Hence, human donor bone procured at the time of death (allografts) and synthetic bone fillers have been used as an alternative to the patient's own bone (autogenous bone graft).

The question that remains is whether additional growth factors that can stimulate bone formation (osteoinductive property) and/or cells that form bone directly (osteogenic property) facilitate healing of these defects when added to a material other than the patient's own bone graft source. In our experience with the use of the synthetic bone graft substitute ultraporous beta-tricalcium phosphate (TCP) (Vitoss, Orthovita, Inc.) over the last 3 years, the graft material, when combined with local blood alone, has performed well clinically but has persisted for a year or longer radiographically in some cases. Prolonged persistence of the graft material may serve as a potential stress riser, although we did not observe any untoward late effects in our published work. Several authors have studied the effects of composite grafts formed from a combination of bone graft substitutes and the patient's own bone marrow in animal models with promising results. There are no studies in the current literature evaluating the effects of healing in composite ultraporous beta-tricalcium phosphate and bone marrow aspirate (BMA) in defects after scraping of benign tumors (cavitary defects) in humans. The purpose of this study is to prospectively examine healing of cavitary defects treated with TCP alone versus those treated with TCP combined with BMA. Our hypothesis is that both graft resorption and trabeculation (radiographic measures of incorporation of the synthetic material by the native bone) will be more advanced at each time point in those patients that receive BMA plus TCP compared to those that receive TCP alone. Patients with any type of benign bone lesion indicated for surgical curettage would be offered inclusion in the study and followed for a minimum of 2 years post-operatively. Bone marrow aspiration would be obtained by a needle inserted through the skin (percutaneous aspiration) from the large bone of the pelvis (iliac crest) using a standard bone marrow aspiration needle. Patients with infection, bone marrow disorders, or other conditions that preclude use of supplementary the patient's bone marrow as well as those who prefer to use their own bone graft material (autograft) or donated human bone graft (allograft) alone would be excluded. Each patient will undergo radiographic evaluation of the lesion at 6 weeks, 3 months, 6 months, 1 year, 18 months and 2 years post operatively. At one time point (1 year) a computerized tomogram (CT) of the grafted region will be obtained for each patient. Two qualified, blinded, independent reviewers will evaluate the radiographs and CT scans for six criteria:

1. presence of graft within the soft tissues,
2. presence of a rim of radiolucency surrounding the grafted defect,
3. size/circumference of the rim of radiolucency,
4. resorption of graft material,
5. trabeculation through the defect and
6. persistence of graft material in the lesion.

Kappa statistics have shown good agreement for these parameters in our retrospective preliminary analysis of results for the TCP use without bone marrow over the first 2 years of its use by the PI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a benign bone lesion requiring surgical curettage

Exclusion Criteria:

* Patients with infection, bone marrow disorders, or other contraindications to use of supplemental bone marrow aspiration as well as those who prefer autologous or allogeneic graft material alone (without synthetic filler) would be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A. Damron, M.D., Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- See also: Paper written in 2002 when study first began — http://www.ncbi.nlm.nih.gov/pubmed/15864061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects seen by Dr. Damron in his clinical office were asked to participate, if they met the inclusion/exclusion criteria. Dates of recruitment February 2005, through August 2007
Groups:
- Vitoss Alone: No bone marrow aspirate used
- Vitoss With Bone Marrow Aspirate: Addition of Vitoss to the bone marrow aspirate
  Vitoss : Synthetic bone graft material
Period: Overall Study
Arm/Group | Vitoss Alone | Vitoss With Bone Marrow Aspirate
Started | 32 | 31
Week 6 Visit | 26 | 28
Month 3 Visit | 25 | 24
Month 6 Visit | 25 | 21
Month 12 Visit | 21 | 25 (Subjects are counted at each milestone as that is when data is collectec)
Month 12 CT Scan | 20 | 25
Month 18 Visit | 21 (As stated previously ea. subject is counted at each milestone, as data is collected at ea. timepoint) | 20
Month 24 Visit | 21 | 18
Completed | 19 | 16
Not Completed | 13 | 15
Not completed — Lost to Follow-up | 6 | 12
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Did not receive vitoss due to infection | 6 | 2

BASELINE CHARACTERISTICS:
Population: Subjects were randomized
Groups:
- Vitoss Used With Bone Marrow Aspirate: Vitoss: Synthetic bone graft material mixed with Bone Marrow aspirate
- Vitoss Only: Vitoss: Synthetic bone graft material alone
- Total: Total of all reporting groups
Arm/Group | Vitoss Used With Bone Marrow Aspirate | Vitoss Only | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 14 | 30
  Between 18 and 65 years | 15 | 17 | 32
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 16 | 17 | 33
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Resorption of Graft Material (GR) Compared at 24 Months
Description: Percentage of graft material that is resorbed (disappears) from area of incorporation, at 24 months .Participants were seen 24 month follow with radiographs to review resorption of graft material. There a several that had incomplete follow up or radiographs not taken.
Time Frame: 24 months
Population: Number of participants analyzed, refers to the number of participants who completed follow up or had radiographs taken at this timepoint.
Measure: Mean (Full Range); unit: percentage of resorption
Groups:
- Vitoss: Addition of Vitoss to the bone marrow aspirate
  Vitoss: Synthetic bone graft material
- Vitoss Alone: Vitoss alone, not bone marrow aspirate used
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 18 | 19
percentage of resorption | 51 [0 to 100] | 47 [0 to 100]
Statistical Analysis 1: Comparison: Vitoss vs Vitoss Alone; The sample size provided at least 80% power at a 5% alpha level to detect a medium to large effect in patients receiving Vitoss alone compared to combination therapy consisting of Vitoss with Bone Marrow Aspirate. Since a random coefficients model was used to analyze the data, the sample size calculation was estimated under this model assuming a 3% attrition rate between all measurement times; Test type: Superiority or Other; p < 0.01, ANOVA; Using baseline (6 wk) and two year post operative predicted effects data, and setting desirable power to detect our effects to 80%

2. Other Pre Specified Outcome: Bone Trabeculation Through the Defect (BT) Compared at 24 Months
Description: Bone trabeculation through the bone lesion at 24 months as determined with radiographs. There were several participants with incomplete follow up or incomplete radiographs. .
Time Frame: 24 months
Population: Number of participants analyzed, refers to the number of participants who completed follow up or had radiographs at this time point.
Measure: Mean (Full Range); unit: percentage of trabeculation
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 18 | 19
percentage of trabeculation | 95 [25 to 100] | 98 [25 to 100]
Statistical Analysis 1: Comparison: Vitoss vs Vitoss Alone; Test type: Superiority or Other; p < 0.01, Chi-squared, Corrected

3. Other Pre Specified Outcome: Resorption of Graft Material (GR) Compared at 18 Months
Description: Percentage of graft material that is resorbed (disappears) from area of incorporation at 18 months. Participants were seen 18 month follow with radiographs to review resorption of graft material. There a several that had incomplete follow up or radiographs not taken.
Time Frame: 18 months
Population: Number of participants analyzed, refers to the number of participants who completed follow up or had radiographs taken at this time point.
Measure: Mean (Full Range); unit: percentage of resorption
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 17 | 17
percentage of resorption | 47 [0 to 100] | 44 [0 to 100]

4. Other Pre Specified Outcome: Bone Trabeculation Through the Defect (BT) Compared at 18 Months
Description: Bone trabeculation through the bone lesion at 18 months with reviewed with radiographs. There were several participants with incomplete follow up or incomplete radiographs.
Time Frame: 18 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage of trabeculation
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 17 | 17
percentage of trabeculation | 90 [25 to 100] | 90 [25 to 100]

5. Other Pre Specified Outcome: Resorption of Graft Material (GR) Compared at 12 Months
Description: Percentage of graft material that is resorbed (disappears) from area of incorporation at 12months. Participants were seen 12 month follow with radiographs to review resorption of graft material. There a several that had incomplete follow up or radiographs not taken.
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage of resorption
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 23 | 19
percentage of resorption | 45 [0 to 100] | 42 [0 to 100]

6. Other Pre Specified Outcome: Bone Trabeculation Through the Defect (BT) Compared at 12 Months
Description: Bone trabeculation through the bone lesion at 12 months was reviewed with radiographs. There were several participants with incomplete follow up or incomplete radiographs.
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage of trabeculation
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 23 | 19
percentage of trabeculation | 42 [25 to 100] | 47 [25 to 100]

7. Other Pre Specified Outcome: Resorption of Graft Material (GR) Compared at 6 Months
Description: Percentage of graft material that is resorbed (disappears) from area of incorporation at 6 months. Participants were seen 6 month follow with radiographs to review resorption of graft material. There a several that had incomplete follow up or radiographs not taken.
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage of resorption
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 19 | 24
percentage of resorption | 28 [0 to 75] | 25 [0 to 75]

8. Other Pre Specified Outcome: Bone Trabeculation Through the Defect (BT) Compared at 6 Months
Description: Bone trabeculation through the bone lesion at 6 months was reviewed with radiographs. There were several participants with incomplete follow up or incomplete radiographs.
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage of trabeculation
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 19 | 24
percentage of trabeculation | 31 [0 to 75] | 33 [0 to 75]

9. Other Pre Specified Outcome: Resorption of Graft Material (GR) Compared at 3 Months
Description: Percentage of graft material that is resorbed (disappears) from area of incorporation at 3 months. Participants were seen 3 month follow with radiographs to review resorption of graft material. There a several that had incomplete follow up or radiographs not taken.
Time Frame: 3 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage of resorption
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 21 | 25
percentage of resorption | 18 [0 to 75] | 22 [0 to 75]

10. Other Pre Specified Outcome: Bone Trabeculation Through the Defect (BT) Compared at 3 Months
Description: Bone trabeculation through the bone lesion compared at 3 months were reviewed with radiographs. There were several participants with incomplete follow up or incomplete radiographs.
Time Frame: 3 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage of trabeculation
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 21 | 25
percentage of trabeculation | 8 [0 to 75] | 10 [0 to 75]

11. Other Pre Specified Outcome: Resorption of Graft Material (GR) Compared at 6 Weeks
Description: Percentage of graft material that is resorbed (disappears) from area of incorporation at 6 weeks. Participants were seen 6 week follow with radiographs to review resorption of graft material. There a several that had incomplete follow up or radiographs not taken.
Time Frame: 6 weeks
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage of resorption
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 27 | 25
percentage of resorption | 6 [0 to 50] | 8 [0 to 50]

12. Other Pre Specified Outcome: Bone Trabeculation Through the Defect (BT) Compared at 6 Weeks
Description: Bone trabeculation through the bone lesion compared at 6 weeks were reviewed with radiographs. There were several participants with incomplete follow up or incomplete radiographs.
Time Frame: 6 weeks
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage of trabeculation
Arm/Group | Vitoss | Vitoss Alone
Number analyzed (Participants) | 27 | 25
percentage of trabeculation | 4 [0 to 50] | 7 [0 to 50]

ADVERSE EVENTS:
Time Frame: 6 week, 3, 6, 12, 18 and 24 months
Description: Subjects were asked at their office visits if they had any new complications, any new diagnosis/treatments, also if records were received from another physician, this information was collected.
Groups:
- Vitoss Without Bone Marrow Aspirate: subjects who received Vitoss without bone marrow aspirate
- Vitoss With Bone Marrow Aspirate: subjects who received Vitoss with bone marrow aspirate
Arm/Group | Vitoss Without Bone Marrow Aspirate | Vitoss With Bone Marrow Aspirate
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 11/32 | 14/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitoss Without Bone Marrow Aspirate (N=32) | Vitoss With Bone Marrow Aspirate (N=31)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Knee pain-persistent (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
recurrence of cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
fracture of wrist (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
bilateral leg weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
drainage at incision (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
femur pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
cervical neuropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
rash at incision (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
fracture of shoulder through lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
fracture of femur through lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitation due to incomplete follow up by subjects or unavailability of radiographs. Also difficulties in assessing the outcomes of resorption if lesions were small or there was artifact from hardware in the area.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No